CLINICAL TRIAL: NCT04146636
Title: Screening in Primary Care of Advanced Liver Fibrosis in NAFLD and/or Alcoholic Patients (IMPROVE Study)
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A01895-52
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: NAFLD; Alcohol-Related Disorder; Liver Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Alcohol-Related Disorders; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: prospective diagnostic study in primary care. Evaluation of a simple blood test (e-LIFT) for the diagnosis of advanced liver fibrosis.
  Reference for advanced liver diagnosis : composite criteria :
  * Elastometry between 8 kPa and 15 kPa and histologic evaluation of fibrosis ≥ F3 (NASH CRN ) OR
  * Elastometry ≥ 15 kPa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic Test: e-LIFT (Other): only one arm because diagnostic study evaluating blood test using elastometry and liver biopsy as reference
  Interventions: Diagnostic Test: e-LIFT

INTERVENTIONS:
Diagnostic Test: e-LIFT — Diagnostic procedure: elastography devices, blood tests (e-LIFT), liver biopsy if necessary (elstometry ≥ 8 kPa and < 15 kPa)

SUMMARY:
The main objective is to determine the performance of the simple eLIFT blood test for advanced liver fibrosis screening in NAFLD and/or alcoholic patients in primary care.

DETAILED DESCRIPTION:
eLIFT, is a new blood fibrosis test specifically dedicated for general practitioners with simple parameters and easy "by head" calculation. Using the recommended cut-offs (eLIFT ≥8), eLIFT sensitivity was 86%. This result position eLIFT an as interesting tool for the screening of advanced liver fibrosis in large populations.

As our preliminary results come from very selected patients, i.e. patients from tertiary centres who underwent a liver biopsy, we now need to evaluate in the real condition of primary care setting whether the use of eLIFT will help general practitioners to screen advanced liver fibrosis in their asymptomatic NAFLD and alcoholic patients.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD and/or alcoholic patient defined by ≥1 of the following criteria:

  * Excessive alcohol consumption: >210 g/week (men), >140 g/week (women)
  * Type 2 diabetes
  * ≥2 metabolic factors among: 1/BMI ≥25kg/m2; 2/elevated blood pressure (antihypertensive drug, or systolic blood pressure ≥130mmHg, or diastolic blood pressure ≥85mmHg), 3/dyslipidemia (lipid-lowering drug, or HDL cholesterol <40mg/dl (men) / <50mg/dl (women), or triglycerides ≥150mg/dl); 4/hyperferritinemia (>300 ng/ml (men)/>200 ng/ml (women))
  * Bright liver at ultrasonography without steatosis-inducing drug
* Obtaining the signature of the consent to participate in the study

Exclusion Criteria:

* Already ongoing specialized follow-up for a chronic liver disease
* Altered health status with poor short-term prognosis, not compatible with a screening procedure
* Decompensated cirrhosis (hepatic encephalopathy, jaundice, ascites, variceal bleeding, hepatorenal syndrome)
* Acute infection
* Inadequate understanding of the French language
* Pregnant, breastfeeding or parturient women
* Persons deprived of their liberty by judicial or administrative decision
* Persons subject to legal protection measures
* Persons unable to consent
* Refusal to participate

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
e-LIFT negative predictive value for the diagnosis of advanced hepatic fibrosis | 1 day
  The primary outcome of the study is the negative predictive value for the diagnosis of advanced hepatic fibrosis (i.e., the rate of patients who do not actually have advanced hepatic fibrosis when the eLIFT test is <8)

SECONDARY OUTCOMES:
sensibility of the eLIFT test | 1 day
  Rate of patients with an eLIFT test ≥8 among patients with advanced hepatic fibrosis
specificity and positive predictive value of the eLIFT test | 1 day
  Rate of patients with an eLIFT test ≥8 but without a final diagnosis of advanced hepatic fibrosis (false positives), specificity (i. e. the rate of patients with an eLIFT test < 8 among patients without advanced hepatic fibrosis) and positive predictive value of the eLIFT test (i. e. the rate of patients with effective advanced hepatic fibrosis when the eLIFT test is ≥ 8)
rate of liver complications among patients with an eLIFT test ≥ 8 | 1 day
  Rate of patients with hepatocellular carcinoma (diagnosed by recommended radiological criteria or liver biopsy); rate of patients with gastroesophageal varices at risk of bleeding diagnosed by gastrointestinal endoscopy (according to Baveno VI rules: medium to large or small varices with red signs) among patients with an eLIFT test is ≥ 8
performance of e-LIFT test in subgroup analysis | 1 day
  Rates of patients with advanced hepatic fibrosis, hepatocellular carcinoma rate, gastroesophageal varicose vein rate at risk of bleeding, eLIFT test rate ≥8, sensitivity, specificity, negative predictive value, positive predictive value in each subgroup (NAFLD, alcohol and NAFLD + alcohol)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Adrien LANNES, Angers, France

IPD SHARING:
Plan to Share IPD: No